CLINICAL TRIAL: NCT03662555
Title: Effect of Neuromuscular Electrical Stimulation Combined With Varying Degrees of Blood Flow Restriction on Muscular and Cardiovascular Function
Brief Title: Effect of Neuromuscular Electrical Stimulation Combined With Blood Flow Restriction on Muscular and Cardiovascular Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Mary's University, Twickenham (Other)
Responsible Party: Principal Investigator, Paul Head, PhD candidate, St. Mary's University, Twickenham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Stmarys
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Muscle Weakness; Muscle Atrophy
MeSH Terms: conditions — Muscle Weakness; Muscular Atrophy | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: In a multi-arm parallel randomised controlled trial design. The randomisation scheme will be generated via online software (http://www.randomization.com). Participants will be recruited to 6 weeks of training, 3 sessions a week and randomised to one of three groups.
  Group 1, participants will undergo NMES and BFR (80% pressure) applied to the quadriceps for 25 min.
  Group 2, participants will undergo NMES and BFR (40% pressure) applied to the quadriceps for 25 min.
  Group 3, participants will undergo NMES alone (Control) applied to the quadriceps for 25 min.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NMES and BFR (80%) (Experimental): Group 1, participants will undergo NMES and BFR (80% pressure) applied to the quadriceps for 25 min.
  Interventions: Device: Neuromuscular electrical stimulation
- NMES and BFR (40%) (Experimental): Group 2, participants will undergo NMES and BFR (40% pressure) applied to the quadriceps for 25 min.
  Interventions: Device: Neuromuscular electrical stimulation
- NMES alone (Active Comparator): Group 3, participants will undergo NMES applied to the quadriceps for 25 min.
  Interventions: Device: Neuromuscular electrical stimulation

INTERVENTIONS:
Device: Neuromuscular electrical stimulation — Neuromuscular electrical simulation (NMES) Two self-adhesive electrodes (2 mm thick) will be placed over the rectus femoris, vastus medialis and vastus lateralis muscles. The electrodes will be placed on the motor points of each muscle. The stimulator discharges biphasic rectangular pulses. The stimulation frequency and duty cycle will be 50 Hz and 5 s of stimulation followed by a 5 s pause for each rep. The intensity of electrical flow will be at each subject's maximum that they can tolerate. The stimulation will be for 5 x 5 min sets with 1 min rest between sets.
  Blood flow restriction
  A handheld Doppler probe (Hi-Dop) will detect their auscultatory and visual pulse using the doppler's screen. The cuff will be inflated initially up to their systolic blood pressure and then incrementally by 10 mmHg until no auscultatory or visual pulse is detected. A percentage of 40% or 80% of each subject's LOP will then be used during the BFR conditions.
  Other Names: Blood flow restriction

SUMMARY:
Neuromuscular electrical stimulation (NMES) has recently been combined with blood flow restriction (BFR) in controlled trials and has shown increased muscular strength and size compared with NMES and BFR on their own. However, none have used BFR pressures previously recommended. The first study of my Ph.D. found 40% and 80% BFR pressures to induce acute fatigue and muscle swelling. However, 80% caused higher ratings of pain and perceived exertion. The present study will determine whether NMES combined with either 40% or 80% BFR causes greater structural muscular adaptations and is perceptually easier after 6 weeks of training.

DETAILED DESCRIPTION:
Laboratory testing will take place on 28 separate occasions, 2 familiarisation, 8 testing and 18 intervention sessions. The first session (FAM 1) will serve as a familiarisation trial to the NMES protocol, BFR stimulus and strength testing. It will be conducted 10-14 days prior to the intervention period. The second session (FAM 2) will serve as a second familiarisation trial to the NMES protocol, BFR stimulus and strength testing. This session will take place 7 days prior to the beginning of the intervention period and will serve as a standardised control period prior to the main testing. The third session (PRE) will take place 1 day prior the start of the intervention period and all future sessions will consist of strength, muscle and cardiovascular function outcome measures. The fourth session (MID) will take place the morning following 3 weeks of training. The fifth session (POST1) will take place 48 hours following 6 weeks of training. There will also be post testing sessions after three days (POST2), one week (POST3) and two weeks post intervention (POST4) to assess detraining. Participants will be provided with protein supplementation after every training session. All strength, muscle and hemodynamic measurements will be conducted at St Marys University by Paul Head. Supplements should be avoided for 72 hours prior to experimental measures and throughout the intervention period. All repeated measures will be performed at a similar time of day (± 1 h).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged between 18 and 45 years old

Exclusion Criteria:

* History of lower extremity surgery, traumatic injuries to the ankle, knee, hip, pelvis and lower back
* Current musculoskeletal condition
* High blood pressure
* Cardiovascular pathology

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-09-26 (Estimated); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Quadriceps volume and muscle architecture (3D Ultrasound) | 8 weeks
  Muscle volume of the vastus lateralis and skeletal muscle architecture will be assessed by ultrasound technique (Telemed LogicScan 128 EXT-1Z). Measurement of fascicle length and pennation angle will be acquired at mid-belly, in the mid-sagittal plane.
Knee extension isometric, eccentric, concentric and endurance strength (Cybex) | 8 weeks
  Maximal isometric, eccentric and concentric strength of the quadricep muscles will be measured using the same isokinetic dynamometer to assess peak force measurements (Cybex). This digital strain gauge dynamometer displays the force measurement to the nearest 0.1 N. Prior to each measurement, the instrument will be calibrated per the manufacturer's instructions and specifications. The individuals will be seated in a comfortable position with the backrest angled at 100˚ to the seat without shoes or orthotic device on. Maximal voluntary isometric contraction (MVIC) for the quadriceps will tested at 60 degrees from full extension using a goniometer (19-21), and the shin pad positioned 2 cm above the lateral malleolus of the fibula attached to a load cell (22).

SECONDARY OUTCOMES:
Voluntary activation | 8 weeks
  The percent of voluntary activation (%VA) will be estimated using the twitch interpolation protocol (25). Doublet stimuli were administered to the femoral nerve approximately 200-300 ms into the MVC. A second doublet will be applied approximately 3 s after the cessation of the MVC at rest (25). The stimuli were rectangular pulses of 200 ls duration and will be delivered using a high-voltage (maximal voltage = 400 V) constant-current stimulator (Digitimer DS7AH, Herthfordshire, UK).
Near-infrared spectroscopy | 8 weeks
  Following 10 min of supine rest a near-infrared spectroscopy (NIRS) optode (Portamon, Artinis medical systems) was placed on the vastus lateralis and secured with an elastic bandage (Tiger Tear, Hampshire, United Kingdom) to prevent movement and covered with an optically dense black material to minimize the intrusion of extraneous light. This protocol was used to characterize the recovery of m˙VO2 and has been shown to be reliable by our group and others (28-30). NIRS will be assessed PRE, MID and POST1, 2, 3 and 4.
Blood pressure | 8 weeks
  A blood pressure cuff (Omron) will be placed around the subject's dominant arm and tested after 5 mins of supine rest and then immediately post each intervention session and at POST testing. To assess acute changes in systolic and diastolic blood pressure. Two readings will be taken and if they have a difference of >5 a third reading will be taken and the average recorded (27).

IPD SHARING:
Plan to Share IPD: No